CLINICAL TRIAL: NCT02086877
Title: COGnitive Outcomes and WELLness in Survivors of Critical Illness
Acronym: COGWELL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, M. Elizabeth Wilcox, Dr. M. Elizabeth Wilcox, University of Toronto
Other Study IDs: 13-6425-BE
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU Survivors who required > 72 hrs mechanical ventilation: No intervention

SUMMARY:
As survival rates from critical illness improve, strategies to return patients to their baseline cognitive and functional status are important research priorities. Up to 100% of ICU survivors will suffer some degree of cognitive impairment at hospital discharge and approximately 50% will have decrements that persist for years. While the mechanisms for this newly acquired brain injury are poorly understood, several risk factors have been identified. Unfortunately, it is unclear how to accurately predict long-term cognitive impairment.

Immediate opportunities to improve cognitive outcomes through risk reduction exist. The investigators propose to comprehensively study the prevalence of sleep abnormalities and their association with cognitive impairment, as it may yield potential targets for effective therapy. Moreover, the investigators will examine for gene x environment associations [APOE ε4] that may allow for genetic risk stratification of individuals at greatest risk of cognitive impairment. The investigators hypothesize that EEG [a sensitive longitudinal marker of brain dysfunction] is a novel and independent predictor of long-term cognitive impairment, and possibly a candidate intermediate end point for future clinical trials.

This study has the potential to identify novel biomarkers and risk factors for post-critical illness cognitive impairment, and may lay the foundation for rational interventions to mitigate risk in high-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years of age
* Admission to study ICU for invasive mechanical ventilation [minimum of 72 hours]

Exclusion Criteria:

* Advanced cognitive impairment or unable to follow simple commands before their acute illness [e.g. end-stage Alzheimer's disease]
* Primary neurological injury [e.g. anoxic brain injury, stroke or traumatic brain injury]
* Anticipated death within 3 months of discharge [e.g. palliative]
* Uncontrolled psychiatric illness at hospital admission
* Not fluent in English
* Unlikely to adhere with follow-up [e.g. no fixed address]
* Residence greater than 300 kms from referral centre

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill individuals who require mechanical ventilation for one week or greater
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance from day 7 after ICU discharge as measured by the Repeatable Battery for the Assessment of Neuropsychological Status [RBANS] and Trail Making Tests A and B | 7 days, 6-months and 12-months after ICU discharge

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form -36 Questionnaire (SF-36) | 7 days, 6- and 12-months after ICU discharge
Beck Depression Inventory-II (BDI-II) | 7 days, 6- and 12-months after ICU discharge
Richard Campbell Sleep Questionnaire | 7 days, 6- and 12-months after ICU discharge
Pittsburgh Sleep Quality Index | 7 days, 6- and 12-months after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: M Elizabeth Wilcox, Principal Investigator — Assistant Professor
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilcox ME, McAndrews MP, Van J, Jackson JC, Pinto R, Black SE, Lim AS, Friedrich JO, Rubenfeld GD. Sleep Fragmentation and Cognitive Trajectories After Critical Illness. Chest. 2021 Jan;159(1):366-381. doi: 10.1016/j.chest.2020.07.036. Epub 2020 Jul 24. PMID 32717265
- [Derived] Wilcox ME, Lim AS, McAndrews MP, Wennberg RA, Pinto RL, Black SE, Walczak KD, Friedrich JO, Taglione MS, Rubenfeld GD. A study protocol for an observational cohort investigating COGnitive outcomes and WELLness in survivors of critical illness: the COGWELL study. BMJ Open. 2017 Jul 13;7(7):e015600. doi: 10.1136/bmjopen-2016-015600. PMID 28710215